CLINICAL TRIAL: NCT05068063
Title: A Randomised Comparison Between Combined Femoral Triangle Block+IPACK Block and Femoral Triangle Block for Anterior Cruciate Ligament Reconstruction Analgesia
Brief Title: Femoral Triangle + IPACK Blocks for ACL Reconstruction Analgesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Chile (Other)
Collaborators: Clinica Alemana de Santiago (Other)
Responsible Party: Principal Investigator, Sebastian Layera, Assistant Professor, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IPACK1
Record Dates: First submitted 2021-09-15; First posted 2021-10-05 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Anterior Cruciate Ligament Rupture; Acute Pain; Pain, Postoperative; Knee Injuries
Keywords: nerve block; IPACK; femoral triangle
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Acute Pain; Pain, Postoperative; Knee Injuries | interventions — Bupivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Femoral Triangle + IPACK block (Experimental): Patients randomized to receive a combination of femoral triangle block and active IPACK block
  Interventions: Drug: Bupivacaine Injection
- Femoral Triangle block (Active Comparator): Patients randomized to receive a combination of femoral triangle block and sham IPACK block
  Interventions: Drug: normal Saline

INTERVENTIONS:
Drug: Bupivacaine Injection — Ultrasound-guided Femoral Triangle block with 20 mL of Bupivacaine 0.25% and IPACK block with 20 mL of Bupivacaine 0.25%
  Arms: Femoral Triangle + IPACK block
Drug: normal Saline — Ultrasound-guided Femoral Triangle block with 20 mL of Bupivacaine 0.25% and IPACK block with 20 mL of normal saline 0.9%
  Arms: Femoral Triangle block

SUMMARY:
An adequate balance between analgesia and motor function is an essential requirement to facilitate functional recovery and early discharge after anterior cruciate ligament (ACL) reconstruction surgery.

Proximal nerve blocks (i.e. femoral and sciatic nerve blocks) are associated with optimal analgesia, but they can cause muscle weakness, interfering with rehabilitation and increasing the risk of falls .

A recent randomized controlled trial concluded that, compared to mid-and distal ACB, a distal femoral triangle block (FTB) is associated with lower opioid consumption and improved postoperative analgesia for ambulatory ACL reconstruction.

In ACL reconstruction surgery there are other potential sources of pain not covered by a FTB, such as intra-articular structures (menisci, cruciate ligaments), posterior knee capsule and the graft donor site.

Evidence supporting the addition of an IPACK block to a FTB has been studied for patients undergoing total knee replacement, nonetheless, there is no trial analyzing the analgesic contribution of IPACK to a FTB in the context of ACL reconstruction surgery.

In this multicentric trial, the investigators set out to analyze the analgesic benefit of adding an IPACK block to a FTB.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled to undergo anterior cruciate ligament reconstruction under general anesthesia with ipsilateral autologous graft.
* Age between 18 and 65 years
* American Society of Anesthesiologists classification 1-3
* Body mass index between 19 and 35 (kg/m2)

Exclusion Criteria:

* Adults who are unable to give their own consent
* Pre-existing neuropathy (assessed by history and physical examination)
* Coagulopathy (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. platelets ≤ 100, International Normalized Ratio ≥ 1.4 or prothrombin time ≥ 50)
* Renal failure (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. creatinine ≥ 100)
* Hepatic failure (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. transaminases ≥ 100)
* Allergy to local anesthetics (LAs), morphine or tramadol
* Pregnancy
* ACL revision surgery
* Contralateral graft or any type of allograft
* Chronic pain syndromes requiring opioid intake at home

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-10-15 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain scores at 2 hours of arrival to Post Anesthesia Care Unit (PACU) | 2 hours after arrival to PACU
  Pain evaluated during knee flexion in Numeric Rating Score from 0 to 10 points

SECONDARY OUTCOMES:
Post-operative static pain scores at 0 hours of arrival to PACU | 0 hours after arrival to PACU
  Pain evaluated at rest in Numeric Rating Score from 0 to 10 points
Post-operative static pain scores at PACU discharge | at discharge of PACU up to 2 hours postoperatively
  Pain evaluated at rest in Numeric Rating Score from 0 to 10 points
Post-operative static pain scores at 6 hours of arrival to PACU | 6 hours after arrival to PACU
  Pain evaluated at rest in Numeric Rating Score from 0 to 10 points
Post-operative static pain scores at 12 hours of arrival to PACU | 12 hours after arrival to PACU
  Pain evaluated at rest in Numeric Rating Score from 0 to 10 points
Post-operative static pain scores at 24 hours of arrival to PACU | 24 hours after arrival to PACU
  Pain evaluated at rest in Numeric Rating Score from 0 to 10 points
Post-operative dynamic pain scores at 0 hours of arrival to PACU | 0 hours after arrival to PACU
  Pain evaluated during knee flexion in Numeric Rating Score from 0 to 10 points
Post-operative dynamic pain scores at PACU discharge | at discharge of PACU up to 2 hours postoperatively
  Pain evaluated during knee flexion in Numeric Rating Score from 0 to 10 points
Post-operative dynamic pain scores at 6 hours of arrival to PACU | 6 hours after arrival to PACU
  Pain evaluated during knee flexion in Numeric Rating Score from 0 to 10 points
Post-operative dynamic pain scores at 12 hours of arrival to PACU | 12 hours after arrival to PACU
  Pain evaluated during knee flexion in Numeric Rating Score from 0 to 10 points
Post-operative dynamic pain scores at 24 hours of arrival to PACU | 24 hours after arrival to PACU
  Pain evaluated during knee flexion in Numeric Rating Score from 0 to 10 points
Femoral Triangle Block success assessment at 2 hours | 2 hours after arrival to PACU
  Sensory block will be assessed with ice on the medial leg
Incidence of opioid related adverse events | 24 hours after arrival to PACU
  Incidence of adverse events related to opioid use (nausea/vomiting, pruritus, somnolence, respiratory depression, urinary retention)
Intraoperative opioid consumption | From anesthesia induction to extubation
  Total opioid use during intraoperative period
PACU opioid consumption | from PACU arrival to discharge up to 2 hours postoperatively
  total opioid consumption during PACU stay
Total opioid consumption | 6 hours, 12 hours and 24 hours after PACU arrival
  Total opioid consumption
Nerve block complications | From nerve block performance up to 24 hours after PACU arrival
  Incidence of nerve block complications (vascular puncture, puncture site erythema, hematoma, foot drop, LAST)
Lower limb tourniquet | from inflation of pneumatic device to tourniquet release
  lower limb tourniquet duration

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Gonzalez, MD, Principal Investigator — Clinica Alemana de Santiago
Locations (2):
- Chile (2):
  - Clinica Alemana de Santiago, Santiago, RM
  - Hospital Clinico Universidad de Chile, Santiago, RM

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wilde J, Bedi A, Altchek DW. Revision anterior cruciate ligament reconstruction. Sports Health. 2014 Nov;6(6):504-18. doi: 10.1177/1941738113500910. PMID 25364483
- [Background] Sharma S, Iorio R, Specht LM, Davies-Lepie S, Healy WL. Complications of femoral nerve block for total knee arthroplasty. Clin Orthop Relat Res. 2010 Jan;468(1):135-40. doi: 10.1007/s11999-009-1025-1. Epub 2009 Aug 13. PMID 19680735
- [Background] Abdallah FW, Whelan DB, Chan VW, Prasad GA, Endersby RV, Theodoropolous J, Oldfield S, Oh J, Brull R. Adductor Canal Block Provides Noninferior Analgesia and Superior Quadriceps Strength Compared with Femoral Nerve Block in Anterior Cruciate Ligament Reconstruction. Anesthesiology. 2016 May;124(5):1053-64. doi: 10.1097/ALN.0000000000001045. PMID 26938989
- [Background] Abdallah FW, Mejia J, Prasad GA, Moga R, Chahal J, Theodoropulos J, Dwyer T, Brull R. Opioid- and Motor-sparing with Proximal, Mid-, and Distal Locations for Adductor Canal Block in Anterior Cruciate Ligament Reconstruction: A Randomized Clinical Trial. Anesthesiology. 2019 Sep;131(3):619-629. doi: 10.1097/ALN.0000000000002817. PMID 31246607
- [Background] Bendtsen TF, Moriggl B, Chan V, Pedersen EM, Borglum J. Redefining the adductor canal block. Reg Anesth Pain Med. 2014 Sep-Oct;39(5):442-3. doi: 10.1097/AAP.0000000000000119. No abstract available. PMID 25140514
- [Background] Johnston DF, Sondekoppam RV, Uppal V, Litchfield R, Giffin R, Ganapathy S. Effect of combining peri-hamstring injection or anterior obturator nerve block on the analgesic efficacy of adductor canal block for anterior cruciate ligament reconstruction: a randomised controlled trial. Br J Anaesth. 2020 Mar;124(3):299-307. doi: 10.1016/j.bja.2019.11.032. Epub 2020 Jan 21. PMID 31980156
- [Background] Johnston DF, Black ND, Cowden R, Turbitt L, Taylor S. Spread of dye injectate in the distal femoral triangle versus the distal adductor canal: a cadaveric study. Reg Anesth Pain Med. 2019 Jan;44(1):39-45. doi: 10.1136/rapm-2018-000002. PMID 30640651
- [Background] Chan E, Howle R, Onwochei D, Desai N. Infiltration between the popliteal artery and the capsule of the knee (IPACK) block in knee surgery: a narrative review. Reg Anesth Pain Med. 2021 Sep;46(9):784-805. doi: 10.1136/rapm-2021-102681. Epub 2021 May 14. PMID 33990439
- [Background] Bushnell BD, Sakryd G, Noonan TJ. Hamstring donor-site block: evaluation of pain control after anterior cruciate ligament reconstruction. Arthroscopy. 2010 Jul;26(7):894-900. doi: 10.1016/j.arthro.2009.11.022. Epub 2010 May 13. PMID 20620788